CLINICAL TRIAL: NCT04594915
Title: Evaluation of Treatment Safety in Patients With Atrial Fibrillation on Edoxaban Therapy in Real-Life in Turkey (ETAF-TR)
Brief Title: Evaluation of Treatment Safety in Patients With Atrial Fibrillation on Edoxaban Therapy in Real-Life in Turkey
Acronym: ETAF-TR
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo Turkey, a Daiichi Sankyo Company (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: ETAF-TR-01
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Atrial Fibrillation
Keywords: Edoxaban; Atrial Fibrillation; Nonvalvular Atrial Fibrillation (NVAF); Non-vitamin K Oral Anticoagulants (NOACs); Real World Evidence (RWE); Turkey
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group: Patients diagnosed with AF who are currently using Edoxaban for stroke prevention in Turkey.
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — Edoxaban according to Package Information (Summary of Product Characteristics [SmPC]).

SUMMARY:
This is a national, multi-center, prospective study to evaluate the safety of Edoxaban in patients diagnosed with AF who are currently using Edoxaban for stroke prevention.

The primary objective:

* To evaluate safety of Edoxaban treatment in patients with atrial fibrillation (AF) on Edoxaban therapy in routine clinical practice in Turkey.

DETAILED DESCRIPTION:
Edoxaban was recently approved by The Turkish Medicines and Medical Devices Agency for the prevention of stroke and systemic embolism in adult patients with Nonvalvular Atrial Fibrillation (NVAF) with one or more risk factors, such as congestive heart failure, hypertension, diabetes mellitus, prior stroke or transient ischemic attack (TIA). Treatment of deep vein thrombosis (DVT) and pulmonary embolism (PE) and prevention of recurrent DVT and PE in adults.

The study will evaluate the safety of Edoxaban in patients diagnosed with AF who are currently on Edoxaban therapy for prevention of stroke in routine clinical practice in Turkey for stroke prevention up to 1 year following treatment by specialized as well as non-specialized physicians in hospital centers.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation (AF) patients aged 18 years or above who are currently using Edoxaban for prevention of stroke.
* Has provided written informed consent to participate in the study.

Exclusion Criteria:

* Not on Edoxaban therapy on the date of obtaining Informed consent
* Receiving Edoxaban therapy for an indication other than the relevant indication (stroke prevention in AF)
* Participating in another ongoing clinical study will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atrial fibrillation patients aged 18 years or above who are currently using Edoxaban for prevention of stroke.
Sampling Method: Non-Probability Sample
Enrollment: 1053 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Number of patients with Overt bleeding following Edoxaban therapy in routine clinical practice in Turkey | From baseline up to 1 year post enrollment
  Overt bleeding is defined as major bleeding or clinically relevant non-major bleeding (CRNM) or any bleeding that does not meet this definition but is considered as overt bleeding by the participating physician. Rates of overt bleeding events will be presented as raw incidence rate (number of patients with events / number of patients treated) and as incidence rates per patient-year (e.g. number of patients with events per 100 patient-years).

SECONDARY OUTCOMES:
Number of Patients with Clinically relevant non-major bleeding following Edoxaban therapy in routine clinical practice in Turkey | From baseline up to 1 year post enrollment
  Rates of clinically relevant non-major bleeding events will be presented as raw incidence rate (number of patients with events / number of patients treated) and as incidence rates per patient-year (e.g. number of patients with events per 100 patient-years).
Number of Patients with Major bleeding following Edoxaban therapy in routine clinical practice in Turkey | From baseline up to 1 year post enrollment
  Rates of major bleeding events will be presented as raw incidence rate (number of patients with events / number of patients treated) and as incidence rates per patient-year (e.g. number of patients with events per 100 patient-years).
Number of Patients with Net Clinical Benefit following Edoxaban therapy in routine clinical practice in Turkey | From baseline up to 1 year post enrollment
  Rates of net clinical benefit will be presented as raw benefit rate (number of patients with benefits / number of patients treated) and as incidence rates per patient-year (e.g. number of patients with events per 100 patient-years).
Number of Patients with Stroke, transient ischemic attack and systemic embolism following Edoxaban therapy in routine clinical practice in Turkey | From baseline up to 1 year post enrollment
  Rates of stroke, transient ischemic attack and systemic embolism events will be presented as raw incidence rate (number of patients with events / number of patients treated) and as incidence rates per patient-year (e.g. number of patients with events per 100 patient-years).
Number of Patients with Major Cardiovascular Events Following Edoxaban Therapy in Routine Clinical Practice in Turkey | From baseline up to 1 year post enrollment
  Rates of major cardiovascular events will be presented as raw incidence rate (number of patients with events / number of patients treated) and as incidence rates per patient-year (e.g. number of patients with events per 100 patient-years).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Daiichi Sankyo Turkey, a Daiichi Sankyo Company
Locations (45):
- Turkey (Türkiye) (45):
  - Başkent University Alanya Practice and Research Hospital, Cardiology Clinic, Antalya, Alanya
  - Ordu University Training and Research Hospital, Ordu, Altinordu
  - Dokuz Eylül University Research and Practice Hospital, Department of Cardiology, Izmir, Balçova
  - Ege University Hospital, Department of Cardiology, Izmir, Bornova
  - Ankara City Hospital, Cardiology Clinic, Ankara, Cankaya
  - Izmir Çiğli Regional Training Hospital, Cardiology Clinic, Izmir, Cigli
  - Aydın Adnan Menderes University Practice and Research Hospital, Department of Cardiology, Aydin, Efeler
  - Private Medinova Hospital, Cardiology Clinic, Aydin, Efeler
  - Istanbul Bezmialem Foundation University, Faculty of Medicine Hospital, Cardiology Clinic, Istanbul, Fatih
  - Health Sciences University Samsun Training and Research Hospital, Cardiology Clinic, Samsun, İlkadım
  - Başkent University İzmir Zübeyde Hanım Practice and Research Hospital, Cardiology Clinic, Izmir, Karsiyaka
  - Medical Park Izmir Hospital, Cardiology Clinic, Izmir, Karsiyaka
  - Muğla Sıtkı Koçman University Training and Research Hospital, Department of Cardiology, Muğla, Mentese
  - Muğla Yücelen Ortaca Hospital, Cardiology Clinic, Muğla, Mentese
  - Balıkesir University Health Practice and Research Hospital, Cardiology Clinic, Balıkesir, Merkez
  - Çanakkale Mehmet Akif Ersoy State Hospital, Cardiology Clinic, Çanakkale, Merkez
  - Çanakkale Onsekiz Mart University Health Application and Research Hospital, Department of Cardiology, Çanakkale, Merkez
  - Tokat Gaziosmanpaşa University, Health Research and Practice Center, Cardiology Department, Tokat Province, Merkez
  - Yozgat City Hospital, Cardiology Clinic, Yozgat, Merkez
  - Bursa City Hospital, Cardiology Clinic, Bursa, Nilüfer
  - Konya Numune Hospital, Cardiology Clinic, Konya, Selcuklu
  - Istanbul Şişli Hamidiye Etfal Training and Research Hospital, Cardiology Clinic, Istanbul, Sisli
  - Eskisehir Umit Private Hospital, Cardiology Clinic, Eskişehir, Tepebaşı
  - Mersin City Training and Research Hospital, Cardiology Clinic, Mersin, Toroslar
  - Van Yüzüncü Yıl University, Dursun Odabaş Medical Center, Van, Tusba
  - Başkent University Istanbul Health Practice and Research Center Hospital, Department of Cardiology, Istanbul, Uskudar
  - Manisa Celal Bayar University Hafsa Sultan Hospital, Department of Cardiology, Manisa, Yunusemre
  - Adana City Training and Research Hospital, Cardiology Clinic, Adana, Yuregir
  - Aksaray Üniversitesi Eğitim Araştırma Hastanesi, Aksaray
  - Ankara Üniversitesi Tıp Fakültesi, Ankara
  - Bayındır Söğütözü Hastanesi, Ankara
  - Medicana International Ankara Hastanesi, Ankara
  - Özel Koru Sincan Hastanesi, Ankara
  - Eskişehir Şehir Hastanesi, Eskişehir
  - Dr. Ersin Arslan Eğitim ve Araştırma Hastanesi, Gaziantep
  - Özel Giresun Ada Hastanesi, Giresun
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi, Istanbul
  - İstanbul Bahçelievler Devlet Hastanesi, Istanbul
  - İstanbul Kartal Koşuyolu Yüksek İhtisas EAH, Istanbul
  - İstanbul Mehmet Akif Ersoy Göğüs Kalp ve Damar Cerrahisi EAH, Istanbul
  - İstanbul Yedikule Göğüs Hastalıkları ve Göğüs Cerrahisi EAH, Istanbul
  - Erciyes Üniversitesi Tıp Fakültesi, Kayseri
  - Manisa Akhisar Mustafa Kirazoğlu Devlet Hastanesi, Manisa
  - Tekirdağ Şehir Hastanesi, Tekirdağ
  - Trabzon Ahi Evren Göğüs Kalp ve Damar Cerrahisi EAH, Trabzon

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Onsel Turk U, Alioglu E, Mavioglu Z, Diker E, Ozpelit E, De Caterina R. Evaluation of Treatment Safety in Patients with Atrial Fibrillation on Edoxaban Therapy in Real-Life in Turkey Study: Design and Rationale. Turk Kardiyol Dern Ars. 2022 Mar 1;50(2):117-123. doi: 10.5543/tkda.2022.21065. PMID 35400633